CLINICAL TRIAL: NCT06559618
Title: A Phase 1B Study to Assess Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Bacteriophage Therapy in Spinal Cord Injury Patients With Bacteriuria
Brief Title: Bacteriophage Therapy in Spinal Cord Injury Patients With Bacteriuria
Acronym: Phage
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Wells Trautner (Other)
Responsible Party: Sponsor-Investigator, Barbara Wells Trautner, Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-54876; 890593 (Other Grant/Funding Number: Craig H. Neilsen Foundation)
Record Dates: First submitted 2024-07-21; First posted 2024-08-19 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Bacteriuria; Spinal Cord Injuries; Asymptomatic Bacteriuria; Escherichia Coli
Keywords: Bacteriophage; Bacteriuria; Phage Therapy; Spinal Cord Injury; Intravesicular infusion; Neurogenic Bladder; Intermittent catheterization; Randomized clinical trial
MeSH Terms: conditions — Bacteriuria; Spinal Cord Injuries; Escherichia coli Infections; Urinary Bladder, Neurogenic | interventions — Phage Therapy

STUDY DESIGN:
Intervention Model Description: Phase 1b, single-center, randomized, double-blind, placebo-controlled study in adults with spinal cord injury with neurogenic bladders and bacteriuria who use indwelling catheters, or who require intermittent catheterization for bladder drainage
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo-controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phage Arm (Experimental): A sterile solution of one to three individual phages (cocktail) (3 x 10^8 plaque forming units [PFU]) phage(s) will be administered intravesicularly (instilled into the participant's bladder via catheter) twice a day for 7 days. The name of the active treatment IP is TAILФR Phage Cocktail (TPC).
  Interventions: Drug: Phage Therapy
- Placebo Arm (Placebo Comparator): Sterile 0.9% saline solution will be instilled into the bladder via catheter twice a day for 7 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Phage Therapy — A 20 mL sterile solution containing one to three individual phage drug substances (TPC) with total strength (potency) 3 x 10^8 plaque-forming units (PFU), will be administered intravesicularly twice a day (one instillation in the morning and one in the evening [at least six hours apart], respectively) for 7 days. The selection of individual phages to include in the TPC are personalized/customized for each participant per phage susceptibility testing to the participant's urinary E. coli (testing is conducted by TAILФR Service Center). Each dose of TPC will be followed with a 10 mL flush of sterile 0.9% saline solution.
  Other Names: Phage
  Arms: Phage Arm
Other: Placebo — Sterile 0.9% saline solution also 20 mL, followed with a 10 mL flush of the same solution.
  Arms: Placebo Arm

SUMMARY:
This is a Phase 1b study to assess the safety, tolerability, PK, and PD of investigational phage therapy (IP) in adults with SCI and bladder colonization (ASB). It is a single-center, randomized, double-blind, placebo-controlled study in adults with SCI with neurogenic bladders and bacteriuria who use indwelling catheters, or who require intermittent catheterization for bladder drainage.

DETAILED DESCRIPTION:
Approximately 30 participants will be randomized 1:1 to receive either investigational phage therapy (3 x 10^8 PFU phage(s)) or inert placebo (sterile normal saline solution) will be administered intravesicularly (instilled into the participant's bladder via catheter) twice a day (BID) for 7 days; the investigational phage therapies are personalized for each participant per phage susceptibility testing to the predominant E. coli pathogen in the participant's bladder. A mixture of up to three phages in a sterile solution will comprise the investigational phage therapy. The study duration for participants will be up to 65 days, which includes up to 30 days for screening, 7 days of IP treatment, and post-treatment assessments at Days 14, 21, 28 and 35 (7, 14, 21 and 28 days after the End of Treatment [EOT] on Day 7, respectively). Day 35 is defined as the EOS. The investigators will strive to enroll participants who are receiving inpatient care in the Spinal Cord Injury units, but enrollment of outpatients with SCI is also possible. Study enrollment will continue for up to 30 evaluable participants.

The study will consist of a Screening Period of up to 30 days. On Day -1, eligible participants will be randomized to investigational phage therapy or placebo. The Treatment Period (Days 1-7) is 7 days and participants will receive a total of 14 doses of IP. The EOT will be after IP dose 14 on Day 7. The Follow-up Period is 35 days starting the day after the EOT with study assessments on Days 14, 21, and Day 35 (EOS). Adverse event data will be collected throughout the study from Treatment Day 1 through the EOS.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Adult (> age 18) inpatients in the SCI care units with neurogenic bladders or outpatients in the SCI care clinics.
4. ASB with E. coli present in a quantity of ≥ 104 CFU/mL).
5. Require an indwelling (transurethral or suprapubic) or intermittent catheterization for bladder drainage.
6. Women of childbearing potential and men with female partners of childbearing potential must use two forms of effective contraception during the study and for two weeks afterwards.
7. Participant will be hospitalized during the 7 days of treatment or will be willing to come into clinic to receive the first dose of IP and training (of participant and/or caregiver) on how to instill the IP into the bladder.

Exclusion Criteria:

1. Unable to provide informed consent for themselves.
2. Received a new antibiotic expected to kill the Gram-negative organisms in the urine between initial enrollment urine culture and the time of randomization.
3. History of neutropenia, defined by ANC < 1000 per µL within 6 months prior to screening.
4. History of organ transplantation.
5. Presence of a surgically-modified bladder, except for a repaired ruptured bladder.
6. HIV with a CD4 count < 200 cells per µL.
7. Unstable vital signs (e.g., fever, hypotension)
8. Symptoms of active urinary tract infection defined as fever, autonomic dysreflexia, generalized increase in spasticity, bladder spasms, new sweating, increase or change in lower abdominal pain, increase in burning or pain when passing urine, increase in burning or pain during catheterization, blood in the urine, or an increased sensation of urinary urgency (MedStar Health, Urinary Symptom Questionnaires for Neurogenic Bladder [USQNB]) (Section 11.2). The presence of any one of these symptoms, unless explained by a non-urinary or non-infectious condition, will be an exclusion criterion.
9. Known urinary obstruction.
10. Medical devices in the urinary tract (other than urinary catheters)
11. Unless deemed acceptable by the sponsor-investigator, prescription drugs, OTC medications and supplements that acidify the urine are excluded.
12. Stage 4 or greater chronic kidney disease
13. Pregnant or breastfeeding female
14. Three or more episodes of autonomic dysreflexia in prior 30 days; defined as those patients who have a SCI and who have had a documented sudden increase in systolic blood pressure of greater than 40 mmHg due to an irritation or stimulation (including bladder or bowel irritation) below the level of the SCI. Autonomic dysreflexia can include findings of hypertensive crisis or emergency, clinically significant bradycardia/tachycardia, severe headache or other severe reaction requiring an acute intervention. The sponsor-investigator will evaluate if a history of severe autonomic dysreflexia is suspected but not clearly identified.
15. In the opinion of the sponsor-investigator, medical or psychiatric illness that would interfere with participation such as active, severe, progressive, or uncontrolled hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, or neurologic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of phage therapy in adults ≥18 years of age with spinal cord injury (SCI) and bacteriuria with Escherichia coli (E. coli) | 2 years
  Safety and tolerability analysis of Adverse Events. The urinary symptom questionnaires provided by MedStar Health, USQNB will be used as a daily study diary.
  Participant's charts for AEs while they are hospitalized, and during study visits on days 14, 21, and 35 if they have been discharged before Day 14.
  Blood samples will be collected for chemistry and hematology on days 1, 3, 7, 14, 21, and 35.
  Urine samples will be collected to detect and analyze markers of inflammation on Days 1, 2, 3, 5, 7, 14, 21, and 35.

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics (PK) of investigational phage therapy | 2 years
  Blood samples will be collected to quantify phage titers, which will be measured as PFU (plaque-forming units) per mL (milliliter) of blood.
  To quantify phage titers, we will perform PCR to measure copies/volume of phage titer compared to a standard control of purified phage.
To evaluate of the pharmacodynamics (PD) of investigational phage therapy | 2 years
  Urine samples will be collected to analyze 1 log reduction in the urinary E. coli on Days 1, 2, 3, 5, 7, 14, 21, and 35.
  Analysis of recurrence of urinary E. coli colonization, incidence of urinary tract infection based on clinical signs and symptoms.
  Microbiological cure, defined as <10^3 CFU/mL of E. coli in the urine on Day 7.

OTHER OUTCOMES:
To explore the influence of phage therapy on the urinary tract microbiota | 2 years
  Urine samples will be collected to analyze microbiome diversity, comparing pre-treatment sample to end of study sample.
  Emergence of phage resistance among the targeted E. coli in the bladder.
To explore the influence of phage therapy on the digestive tract microbiota | 2 years
  Analysis of stool sample microbiome diversity, comparing pre-treatment to end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara W Trautner, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Terwilliger A, Clark J, Karris M, Hernandez-Santos H, Green S, Aslam S, Maresso A. Phage Therapy Related Microbial Succession Associated with Successful Clinical Outcome for a Recurrent Urinary Tract Infection. Viruses. 2021 Oct 12;13(10):2049. doi: 10.3390/v13102049. PMID 34696479
- [Background] Green SI, Kaelber JT, Ma L, Trautner BW, Ramig RF, Maresso AW. Bacteriophages from ExPEC Reservoirs Kill Pandemic Multidrug-Resistant Strains of Clonal Group ST131 in Animal Models of Bacteremia. Sci Rep. 2017 Apr 12;7:46151. doi: 10.1038/srep46151. PMID 28401893
- [Background] Salazar KC, Ma L, Green SI, Zulk JJ, Trautner BW, Ramig RF, Clark JR, Terwilliger AL, Maresso AW. Antiviral Resistance and Phage Counter Adaptation to Antibiotic-Resistant Extraintestinal Pathogenic Escherichia coli. mBio. 2021 Apr 27;12(2):e00211-21. doi: 10.1128/mBio.00211-21. PMID 33906920
- [Background] Green SI, Clark JR, Santos HH, Weesner KE, Salazar KC, Aslam S, Campbell JW, Doernberg SB, Blodget E, Morris MI, Suh GA, Obeid K, Silveira FP, Filippov AA, Whiteson KL, Trautner BW, Terwilliger AL, Maresso A. A Retrospective, Observational Study of 12 Cases of Expanded-Access Customized Phage Therapy: Production, Characteristics, and Clinical Outcomes. Clin Infect Dis. 2023 Oct 13;77(8):1079-1091. doi: 10.1093/cid/ciad335. PMID 37279523